CLINICAL TRIAL: NCT00777075
Title: Oral Administration of L-Arginine in Patients With Erectile Dysfunction
Brief Title: L-Arginine and Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: Pharmacia (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B VP2.A-7140-00-37/4020796
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2008-10-22 (Estimated); Status verified 2008-10

CONDITIONS: Erectile Dysfunction
Keywords: nitrate; nitric oxide; asymmetric dimethylarginine; blood pressure; NOS; IIEF
MeSH Terms: conditions — Erectile Dysfunction | interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-arginine (Active Comparator)
  Interventions: Drug: L-arginine
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-arginine
  Arms: L-arginine
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of the study is to determine whether the treatment with L-arginine leads to an improvement of erectile dysfunction in patients with erectile dysfunction.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is a common medical disorder often affecting the aging male. Nitric oxide (NO) is a physiological signal essential to penile erection. NO synthase (NOS) catalyzes the production of NO from L-arginine. ADMA, a competitive inhibitor of NO synthase increases with age and many disorders that reduce NO in the erectile tissue are commonly associated with ED. Although new pharmacological strategies have been identified for medical treatment of ED, patients often seek alternative therapies for cost or side effect reasons.

The aim of the present study is to determine the efficacy of orally administered L-arginine on ED not caused by established organic disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 20 and 65 years, an ED for at least 6 months duration and written consent.
* Each patient had to be informed about the study details in written and oral form before the beginning of the drug administration.
* The hormonal status including dehydroepiandrosterone sulfate (DHEAS), Prolactin and Testosteron of each patient had to be within the normal range. -

Exclusion Criteria:

* Patients with primary erectile dysfunction, congenital anomalies, Diabetes mellitus, severe hepatic-and renal insufficiency, severe cardiovascular diseases, cerebrovascular accidents, uncontrolled hypertension, endocrine diseases, psychiatric disorders, and evidence of dementia were excluded.
* Patients were excluded if they had pelvic fractures or prostatectomy and if they had undergone reconstructive or prosthetic surgery on the penis.
* Increased levels of serum potassium, known hypersensitivity to the study medication or any ingredient of the drug.
* Administration of PDE-5-Inhibitors (sildenafil, tadalafil, vardenafil or apomorphine) within four weeks prior to the administration of l-arginine or placebo led to exclusion.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57
Dates: Start 2003-07; Study Completion 2005-11

PRIMARY OUTCOMES:
International Index of Erectile Dysfunction | 16 weeks

SECONDARY OUTCOMES:
L-arginine plasma-levels | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dirk O. Stichtenoth, MD, Study Director — Institute of Clinical Pharmacology, Hannover Medical School
Locations (1):
- Institute of Clinical Pharmacology, Hannover Medical School, Hanover, Lower Saxony, Germany